CLINICAL TRIAL: NCT04513678
Title: Development of ImmunOncoTool: A Web-Based irAE Monitoring Platform
Brief Title: Development of ImmunOncoTool
Acronym: ACS-MRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Cancer Society, Inc. (Other); Bristol-Myers Squibb (Industry); Melanoma Research Foundation Breakthrough Consortium (Other)
Responsible Party: Principal Investigator, Betina Yanez, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00207560
Record Dates: First submitted 2020-08-07; First posted 2020-08-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Cancer; Cancer, Treatment-Related
Keywords: eHealth; Symptom Burden; Health Related Quality of Life; Immunotherapy
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImmunOncoTool Condition (Experimental): The ImmunOncoTool condition includes access to the web-based platform, routine monitoring of irAEs every week for twelve weeks and then bi-weekly for an additional eight weeks, and messages to healthcare providers and patients if a reported irAE is deemed severe enough that it warrants provider attention.
  Interventions: Behavioral: ImmunOncoTool Condition
- Control (No Intervention): Participants in the control condition are not assigned an intervention. They receive standard of care.

INTERVENTIONS:
Behavioral: ImmunOncoTool Condition — Immunotherapy education + irAE monitoring + Facilitation of patient-provider communication
  Other Names: Experimental
  Arms: ImmunOncoTool Condition

SUMMARY:
The purpose of this study is to facilitate the recognition and early management of Immune Related Adverse Events (irAEs) experienced by cancer patients taking immunotherapy. This is done through the development of a web-based platform in which patients receive valuable education about irAEs, patients' irAEs are routinely monitored, patient reported irAEs are embedded into patient clinical care, and patient-provider communication and prompt management of irAEs is facilitated.

The intervention component includes access to the web-based platform, routine monitoring of irAEs every week for twelve weeks and then bi-weekly for an additional eight weeks, and messages to healthcare providers and patients if a reported irAE is deemed severe enough that it warrants provider attention.

Participants are randomized into either an intervention group (described above) or a control group, in which their irAEs are monitored once after a twelve week interval and again after an additional eight weeks. Additionally, both intervention and control participants complete three assessments: baseline (at the beginning of the research study), 12-week follow-up, and 20-week follow-up.

DETAILED DESCRIPTION:
Experiencing adverse events can compromise the clinical benefit of a cancer treatment, and may go undetected by clinicians. Specific to checkpoint inhibitors, Immune Related Adverse Events (irAEs) include symptoms such as fatigue, headaches, skin reactions, nausea or vomiting, diarrhea as well as colitis, liver toxicities, and endocrinopathies. A systematic review for 50 clinical trials with a total of 5,071 patients receiving immune checkpoint inhibitors revealed that grade 3 or 4 irAEs were present in up to 66% of patients. In general, if irAEs are detected quickly, they are reversible and manageable with immunosuppressive therapy. However, severe or life-threatening irAEs may lead to discontinuation of the checkpoint inhibitor, which can lead to cancer progression and ultimately patient mortality. Therefore, prompt recognition and management of irAEs before they become severe can prevent irAEs that may be life-threatening as well as prevent discontinuation of checkpoint inhibitors.

Web-based interventions provide flexibility and overcome many obstacles to accessibility for patients who may not be able to meet at a certain location due to disease-related physical limitations or logistical limitations. Specific to cancer, web-based interventions have demonstrated efficacy in reducing depressive symptoms, distress, and improved functional well-being among patients with cancer. Finally, web based platforms are useful for monitoring patient-reported outcomes and linking outcomes to providers. Overall, web-based monitoring and embedding of patient-reported adverse events into clinical care can improve cancer outcomes. To the best of our knowledge, no study has established the efficacy of a platform that links patient-reported irAEs to oncology providers.

Our primary outcome will measure the feasibility of the digital health program, ImmunOncoTool. Our secondary outcome will be the preliminary intended effects of ImmunOncoTool which will be assessed through endpoints such as clinician response and time to clinician response of patient-reported irAEs, number and length of unscheduled breaks in checkpoint inhibitor treatment and discontinuation of checkpoint inhibitor treatment, length of time spent managing any irAEs, provider reported irAEs, and concurrence between patientreported irAE and provider reported irAEs as these factors may explain the effect of ImmunOncoTool on improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Provider and electronic medical report (EMR) confirmed diagnosis of lung, kidney, urothelial, or melanoma cancer as checkpoint inhibitors are used primarily in these disease sites
* English-speaking as the content and website will only be available in English for feasibility testing
* Have initiated a checkpoint inhibitor
* Have access to the internet

Exclusion Criteria:

* significant cognitive impairment or inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis)
* concurrent cancer-related treatment aside from checkpoint inhibitors
* pre-existing auto-immune condition which may impact the course of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Demand of ImmunOncoTool: Recruitment Rate | 20 weeks
  We assess demand of the ImmunOncoTool application through study recruitment. Based on previous psychosocial and behavioral studies in oncology, an 80% recruitment rate is considered an adequate level of demand.
Demand of ImmunOncoTool: Retention Rate | 20 weeks
  Another way we assess demand of the ImmunOncoTool application is through participant retention. Based on previous psychosocial and behavioral studies in oncology, an 80% retention rate is considered an adequate level of demand.
Acceptability of ImmunOncoTool | T2 (immediately following 12 week intervention)
  To assess acceptability, all participants are asked to complete an exit interview on ImmunOncoTool. This interview assesses usefulness, satisfaction, learnability and usability of the application. This exit interview was synthesized from validated measures assessing eHealth intervention feasibility, and was adapted for our study to better fit our target population and our application design. Above average scores on the questionnaire are considered acceptable. The satisfaction questionnaire is administered over the phone immediately following the 12 week intervention.
Engagement of ImmunOncoTool: Number of Login's | 20 weeks
  We assess engagement of the ImmunOncoTool application by examining the number of participant logins to the web-based application.
Engagement of ImmunOncoTool: Duration of Usage | 20 weeks
  We assess engagement of the ImmunOncoTool application by examining the duration participant time spent on the website. Based on previous psychosocial and behavioral studies in oncology, an average of 8 hours of use is considered an adequate level of engagement.
Engagement of ImmunOncoTool: Content Accessed | 20 weeks
  We assess engagement of the ImmunOncoTool application by examining the type of content accessed by participants on the website.

SECONDARY OUTCOMES:
Change in Health Related Quality of Life will be evaluated with The Functional Assessment of Cancer Therapy (FACT-G8) | T1 (prior to starting intervention), T2 (immediately following 12 week intervention), T3 (2 months following intervention)
  The FACT-G8 is a validated questionnaire that assesses top-rated symptoms and concerns for a broad spectrum of advanced cancers and serves as a health-related quality of life (HRQoL) measure.
Healthcare Utilization Form | T2 (immediately following 12 week intervention), T3 (2 months following intervention)
  The Healthcare Utilization Form is used in order to capture possible medical events outside of the NU system that research staff was not able to catch through the patients' electronic medical record.
Immune Related Adverse Events (irAEs) are measured with the Health Questionnaire. | T1 (prior to starting intervention), every week during the 12 week intervention, T2 (immediately following 12 week intervention), biweekly for 8 weeks immediately following intervention, T3 (2 months following intervention)
  The Health Questionnaire assesses the severity of symptoms patients may feel that often correspond with immunotherapy. These symptoms can provide information regarding possible irAEs experienced by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Betina Yanez, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with any researchers outside Northwestern.

DOCUMENTS (1):
  • Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT04513678/ICF_000.pdf